CLINICAL TRIAL: NCT07088705
Title: Pioneering Verification of the Use of the Immunomodulatory Effect of Subthreshold Micropulse Laser Therapy (SML) in Retinitis Pigmentosa With an Attempt to Optimize 577 nm and 810 nm Laser Protocols
Brief Title: Subthreshold Micropulse Laser Therapy (SML) in Retinitis Pigmentosa
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Marta P. Wiącek (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor-Investigator, Marta P. Wiącek, PhD, Pomeranian Medical University Szczecin
Organization: Pomeranian Medical University Szczecin (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/ABM/03/00014
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Retinitis Pigmentosa (RP)
Keywords: Retinitis Pigmentosa; subtreshold micropulse laser; treatment
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SML 577 nm (Experimental): Patient preparation will include obtaining informed consent, local anesthesia of the conjunctival sac with 0.05% proxymetacaine drops to reduce discomfort, and the administration of 0.1% tropicamide to dilate the pupil and increase access to the retina during laser stimulation. Next, a Volk macular contact lens (Volk Optical, Mentor, OH, USA) will be placed on the cornea using a viscoelastic agent. A modern 577 nm yellow laser (Supra Scan 577, Quantel Medical, Cedex, France) will be used for stimulation. The panmacular stimulation is planned, with the laser covering the entire central retinal area between the vascular arches, including the foveal region. Approximately 600 160-μm diameter impacts will be delivered per session using a 250-μm power output with a duration of 0.2 seconds and a 5% duty cycle.
  Interventions: Device: SML 577 nm
- SML 810 nm (Active Comparator): Preparation for SML using an 810 nm red laser will involve informed consent, local anesthesia of the conjunctival sac with 0.05% proxymetacaine drops to reduce discomfort during the procedure, and the administration of 0.1% tropicamide to dilate the pupil and increase access to the retina during laser stimulation. A Volk macular contact lens (Volk Optical, Mentor, OH, USA) will then be placed on the cornea using a viscoelastic agent. Central retinal stimulation will be performed using an 810 nm SML. The panmacular stimulation protocol will be used, with the laser covering the entire central retinal area between the vascular arcs, including the foveal region. During one session, approximately 1500-2000 confluent local applications of 200 μm diameter will be performed using 1.4 W of power with a duration of 0.15 seconds and a 5% duty cycle.
  Interventions: Device: SML 810 nm
- Sham SML (Sham Comparator): It is worth emphasizing that the experiment was designed as a factorial study design with the patient blinded. To this end, patient preparation, laser treatment duration, and auditory and visual sensations during the sham procedure will be the same as those experienced with a truly lasered eye. Consequently, fellow eye of an each RP eye that undergone the SML stimulation in either arm 1 or 2 will be included in the sham group (60 eyes).
  Interventions: Other: Sham SML

INTERVENTIONS:
Device: SML 577 nm — A 577 nm yellow and 810 nm red lasers will be used for stimulation. The panmacular stimulation is planned, with the laser covering the entire central retina between the vascular arches, including the foveal region according to the study protocol.
  Patient preparation will include obtaining informed consent, local anesthesia of the conjunctival sac with 0.05% proxymetacaine drops to reduce discomfort, and the administration of 0.1% tropicamide to dilate the pupil and increase access to the retina during laser stimulation. Next, a Volk macular contact lens (Volk Optical, Mentor, OH, USA) will be placed on the cornea using a viscoelastic agent. A modern 577 nm yellow laser (Supra Scan 577, Quantel Medical, Cedex, France) will be used for stimulation. The panmacular stimulation is planned, with the laser covering the entire central retinal area between the vascular arches, including the foveal region.
  Arms: SML 577 nm
Device: SML 810 nm — Preparation for SML using an 810 nm red laser will involve informed consent, local anesthesia of the conjunctival sac with 0.05% proxymetacaine drops to reduce discomfort during the procedure, and the administration of 0.1% tropicamide to dilate the pupil and increase access to the retina during laser stimulation. A Volk macular contact lens (Volk Optical, Mentor, OH, USA) will then be placed on the cornea using a viscoelastic agent. Central retinal stimulation will be performed using an 810 nm SML. The panmacular stimulation protocol will be used, with the laser covering the entire central retinal area between the vascular arcs, including the foveal region. During one session, approximately 1500-2000 confluent local applications of 200 μm diameter will be performed using 1.4 W of power with a duration of 0.15 seconds and a 5% duty cycle.
  Arms: SML 810 nm
Other: Sham SML — It is worth emphasizing that the experiment was designed as a factorial study design with the patient blinded. To this end, patient preparation, laser treatment duration, and auditory and visual sensations during the sham procedure will be the same as those experienced with a truly lasered eye. Consequently, fellow eye of an each RP eye that undergone the SML stimulation in either arm 1 or 2 will be included in the sham group (60 eyes).
  Arms: Sham SML

SUMMARY:
Introduction Retinitis pigmentosa (RP) is the most common form of genetic retinal degenerative disease. The disease is progressive and leads to blindness and permanent disability within a few years of diagnosis. The etiology of RP is multifactorial. It combines genetic (multiple inheritance patterns) and environmental factors, which makes it difficult to develop effective causal therapy. Many potential methods of RP treatment have been described so far, but the lack of unequivocal evidence of the therapeutic effectiveness of these methods implies a lack of RP therapy standards. Few analyzes have shown that the use of a red subthreshold micropulse laser (SML) with a wavelength of 810 nm causes a neurostimulatory effect on the retina. The subsequent introduction of a yellow laser with a wavelength of 577 nm, dedicated to edema and ischemic retinal diseases, re-initiated a series of questions about the effectiveness of both therapies and the treatment protocols used. This fact emphasizes the need for further verification and optimization of SML treatment regimens in Poland, which has a chance to become a new, widely available, non-invasive standard of treatment independent of the genetic pattern.

The aim of the project The main goal of the experiment is to verify the effectiveness of SML and determine the optimal treatment protocol for SML based on a detailed analysis of molecular changes of selected pro-inflammatory, neurotrophic and angiogenic factors (IL-1α, IL-1β, IL-2, IL-4, IL-5, IL- 6 IL-8, IL-10, IL-12 p70, IL-13, IL-17A, CXCL8 / IL-8, MCP-1 / CCL2, MIP-1α / CCL3, MIP-1β / CCL4, IL-8 / CXCL8, CCL5 / RANTES, IP-10 / CXCL10, GM-CSF, MMP-2, MMP-3, MMP-7, MMP-8, MMP-9, MMP-13, BMP-4, BMP-7, BMP - 9, TIMP-1, t-PA, PAI-1, NGF, EGF, TNF-α, TGF-β1, TGF-β2, FGF, EGF, G-CSF, GM-CSF, HGF, PDGF-AA, PDGF- AB / BB, VEGF, PAI-1, COL1A1, TSP-2, IFN-γ, N-cadherin, E-selection and P-selection) in tears and peripheral blood of patients with RP. Moreover, the project aims to personalize the assessed treatment regimens by determining the correlation between these changes and the genotype and dynamics of functional changes of the retina in the eyes from the RP subjected to single stimulation with yellow and red SML.

Materials and methods The study group will consist of 60 adult patients with retinitis pigmentosa diagnosed on the basis of a characteristic clinical picture confirmed by genome analysis using the whole exome sequencing method and full-field electroretinoography (ERG). In randomized selection, one eye of each patient will be randomly assigned to be stimulated with red (30 eyes) or yellow (30 eyes) SML, and second eye will be assigned to the sham procedure. This will ensure a comprehensive comparative assessment of the effectiveness of both types of SML against each other and against a placebo. The tear film will be collected by wetting the Schirmer strips placed under the lower eyelid before SML (T0) and 28 days (T1), 3 months (T2) and 6 months (T3) after the laser stimulation. In addition, approximately 7.5 ml of peripheral venous blood will be collected at corresponding time points. The assessment of the dynamics of functional changes based on the measurements of the best corrected visual acuity for distance and near vision, contrast sensitivity, microperimetry, 10-2 and 30-2 static perimetry, electroretinogram stimulated with the pattern (PERG) and multifocal electroretinogram (mfERG) in both eyes will be carried out at the time points T0, T1-T3. In addition, during the T0-T3 visits, the morphology of the eyeball, i.e. examination of the anterior segment and fundus of the eye in a slit lamp, examination of optical coherence tomography of the macula and ultrasound of the eyeball will be assessed. The quality of life of the participants of the experiment will be assessed on the basis of the standardized NEI VFQ-25 questionnaire. The quality of life assessment will take place both before the implementation of the SML and during subsequent follow-up visits.

Expected project benefits Conducting the proposed experiment will result in verification of the effectiveness of the retinal stimulation by the yellow SML in comparison to the red SML in the eyes with retinitis pigmentosa. In addition, conducting genome analysis and monitoring changes in the concentration of pro-inflammatory, neurotrophic and angiogenic factors in the tear film and peripheral blood in combination with a detailed assessment of the dynamics of functional changes in the eyes with RP after stimulation with an immunomodulatory stimulus SML will enable optimization and personalization of this treatment method in relation to the genetic profile of the patient with RP. The expected results may direct further research on the search for an effective therapy for patients with RP or constitute the basis for the introduction of the world's first standard of adjuvant treatment in this disease entity.

DETAILED DESCRIPTION:
It is estimated that there are approximately 10,000 patients with RP in Poland. Taking into account the inclusion criteria, recruitment duration, the specificity and innovative nature of the experiment, and logistical constraints, the investigators planned to recruit 60 adult patients with RP who met both the inclusion and exclusion criteria. The diagnosis of RP will be made based on the characteristic clinical picture: (i) a typical RP fundus appearance with a waxy pallor of the optic disc; (ii) reduced retinal vessel diameter and intraretinal pigment deposits in the central periphery of the fundus; (iii) a history of progressive night and/or color vision impairment, peripheral vision loss, photophobia, reduced visual acuity, and prolonged dark adaptation; (iv) peripheral narrowing, even to "tunnel vision" on visual field testing. Additionally, to confirm the diagnosis, Next-Generation Sequencing (NGS) will be performed, covering all known genes responsible for retinal dystrophic diseases, or genome analysis using whole exome sequencing (WES). Furthermore, each patient will undergo full-field electroretinography (ERG), where the expected result for RP indicates a significant reduction or inability to detect a response from the peripheral retina. It is worth emphasizing that appropriate selection criteria, combined with the pioneering combination of a detailed functional and morphological assessment of the eyeball subjected to SML and cytogenetic analysis, could represent a breakthrough in the search for the first effective standard of treatment for RP.

It is noteworthy that the diagnosis is usually made in the 2nd or 3rd decade of life, the gradual progression of visual impairment with predicted vision loss, and the lack of effective treatment options make the diagnosis of RP emotionally devastating. This disease is progressive, leading to progressive blindness and permanent disability within a few years of diagnosis. This poses a significant problem for patients, their caregivers, the healthcare system, and society as a whole. Furthermore, the inability to independently perform previously achievable activities and dependence on others lead to frustration and low self-confidence, leading to life dissatisfaction and depressive symptoms. Consequently, patients with RP experience decreased motivation to perform daily tasks, including work, which ultimately burdens the social and welfare system. On the other hand, the progressive nature of RP forces patients to constantly adapt to daily challenges, which become increasingly difficult due to deteriorating visual function. The deteriorating quality of life scores in patients with RP, depending on disease progression, indicate that visual replacement skills may not be sufficient to cope with social interactions in the advanced stages of the disease. This condition is currently incurable due to the lack of causal therapy. Moreover, due to the multifactorial nature of the condition, including a combination of environmental and genetic factors, developing causal treatments for RP is an extremely difficult challenge. Furthermore, there is currently no effective symptomatic therapy to inhibit disease progression. Therefore, there is an urgent need to find effective treatment methods and correlate treatment response with phenotypic and genotypic conditions, also in the Polish population. The use of the increasingly widely available, inexpensive method of non-invasive retinal stimulation using SML to induce immunomodulatory and regenerative effects on damaged photoreceptors raises hopes for the first effective treatment to inhibit disease progression in RP.

There are only few reports in the medical literature on the relationship between the severity of retinal degeneration in the RP and disturbed expression of microglia and proinflammatory cytokines. However, no detailed analysis of this issue, especially in the context of the genetic profile, as well as its potential use in the development of therapeutic methods of the RP has been carried out. The introduction of SML to the treatment of retinal diseases has revolutionized the way laser therapy is perceived in ophthalmology. During SML, laser energy is delivered to the retinal pigment epithelium (RPE) in the form of a series of very short pulses, between which there are pauses to allow the tissue to cool down, so no damage to the cells is caused. It has been shown that this energy activates the heat shock proteins in RPE. The mode of action of these proteins is based on their anti-inflammatory and anti-angiogenic effects and cause the local increase in cytokine concentration which leads to the induction of acute inflammation. The consequence of this condition, caused by the induction of an immunomodulatory effect, is the reduction of the chronic inflammation responsible for the formation of degenerative changes in the retina. Moreover, the process of protein secretion by the RPE optimizes and improves functioning of the retina. This mechanism may be important especially in degenerative diseases of the retina, where there is a progressive impairment of the RPE function. It is worth emphasizing that this method is not associated with the risk of permanent damage to the retina and no side effects have been described so far. In the world literature, only two analyzes of the effectiveness of the red SML stimulus in the eyes from RP have been reported so far, showing significant benefits in terms of improving visual acuity, visual field and function of the retinal ganglion cells. It should be noted, however, that this material concerned a retrospective evaluation with a short observation period of 1 month and was carried out on a limited number of patients. Additionally, the selection of diagnostic methods did not provide a complete assessment of the dynamics of functional changes in the retina. Moreover, it seems that such a short time of observation of patients does not allow to differentiate the short-term effect of the applied therapy and the physiological fluctuations in the parameters of the organ of vision in the course of RP. Importantly, no study using the innovative yellow SML stimulus in the panmacular protocol in the eyes of the polish inhabitants has been published so far. In conclusion, the available material is too limited to define the effect of the SML stimulus on immunomodulatory processes and define SML as a recommended treatment procedure for RP.

The planned medical experiment is the first comparison of the neurostimulatory effects of two SMLs on the RP, of which one (red) has already shown some efficacy in this disease entity, but there is no agreement between researchers as to the optimal retinal laser protocol. The second laser (yellow) is, in turn, a representative of the new generation of these devices with a shorter wavelength, which may increase the safety of the procedure with the simultaneous intensification of action in the area of the damaged retina. Additionally, the innovative nature of the project is supported by the fact that it will be the first experiment to determine the cytogenetic profile in patients with RP in combination with the evaluation of the modulation of proinflammatory, neurotrophic and angiogenic factors in tears and peripheral blood as well as functional changes of the eyeball in the course of using both SML.

The meticulous study protocol was provided in corresponding sections of the clinical trial registration form.

ELIGIBILITY:
Inclusion criteria:

* Clinically diagnosed RP, including (i) characteristic fundus appearance with waxy pallor of the optic disc; (ii) reduced retinal vessel diameter and intraretinal pigment deposits in the central periphery of the fundus; (iii) history of progressive night vision and/or color vision impairment, peripheral vision loss, photophobia, reduced visual acuity, and prolonged dark adaptation; (iv) peripheral narrowing to "tunnel vision" on visual field testing; (v) significant amplitude reduction with prolonged waveform latency or unrecordable readings on flash electroretinography (ERG) and confirmed by NGS panel sequencing covering all known genes responsible for retinal dystrophic diseases or Whole Exome Sequencing (WES);
* Age 18-70 years; - BCDVA no lower than 0.08 (according to the Snellen chart);
* Ability to provide informed consent.

Exclusion criteria:

* Age <18 years - >70 years;
* Systemic diseases (acute inflammatory or autoimmune process, recent trauma, renal or hepatic failure, cardiovascular or neurological disease, stroke, cancer, diabetes, autoimmune diseases);
* Other eye diseases (e.g., glaucoma, age-related macular degeneration, vitreous degeneration); - Post-ocular surgery except uncomplicated cataract surgery;
* Cataract surgery or posterior capsulotomy less than 3 months prior to study enrollment;
* Systemic or topical use of immunomodulatory medications;
* Use of any other RP treatment, including dietary supplements, during the study or in the 3 months prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
BCDVA improvement | The planned follow-up time is 6 months with visits before the intervention, at 1, 3 and 6 months after the SML procedure.
  BCDVA improvement is defined as an increase of at least 5 letters demonstrated at at least two consecutive time points after the intervention compared to baseline measurements. BCDVA is visual acuity measured using standardized ETDRS charts, measuring the number of letters read correctly by the patient at a distance of 4 meters.

SECONDARY OUTCOMES:
Improvement in the bioelectrical function of the central retina assessed by mfERG. | The planned follow-up time is 6 months with visits before the intervention, at 1, 3 and 6 months after the SML procedure.
  The bioelectrical function of the cone system and bipolar cells will be recorded in the mfERG test according to the widely recognized standards of the International Society for Clinical Electrophysiology of Vision (ISCEV). Improvement in the bioelectrical function of the central retina assessed by mfERG will be determined based on analysis of the P1 wave amplitude from the central 60° angle, presented separately for six concentric rings. Furthermore, the result will be interpreted as a P1 wave response map generated after stimulation of the central retina by pseudorandomly displaying hexagonal fields with standardized, high contrast on a special computer monitor while maintaining visual fixation. This recording is performed under daytime adaptation conditions.
The improvement of mean deviation (MD) in 10-2 perimetry. | The planned follow-up time is 6 months with visits before the intervention, at 1, 3 and 6 months after the SML procedure.
  The main complaint of patients with RP and a parameter enabling the assessment of the severity and rate of disease progression is visual field testing with the assessment of mean deviation (MD) in perimetry. Due to the usually significant loss of peripheral photoreceptors, a more sensitive test is the 10-2 protocol with the assessment of central retinal sensitivity compared to broader measurements, including those performed 24-2 as a screening test for various disease entities.
Improvement of a macular integrity and retinal sensitivity in a microperimetry test | The planned follow-up time is 6 months with visits before the intervention, at 1, 3 and 6 months after the SML procedure.
  Measuring macular integrity and retinal sensitivity in a modern microperimetry test is a test that determines retinal sensitivity in various foveal and perifoveal areas. It is a functional assessment technique that provides a direct correlation between anatomical and functional findings.

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Ophthalmology, Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Yes
No personal data that could be used to identify precisely what individuals were enrolled for the study can be revealed. However, all clinical data including ophthalmic measurements might be available on a request.
Supporting Information: Study Protocol
Time Frame: The data will be available as soon as they will be acquired (August 2026) for at least 10 consecutive years.
Access Criteria: The data will be available on a request directed to the principal investigator of the study. Especially the publishing journal and researchers planning to perform further analysis involving the study data are authorized.